CLINICAL TRIAL: NCT03900000
Title: Improved Orthostatic Tolerance = Better Cognitive Function in Parkinson's Disease: Does a Successful Treatment of Orthostatic Hypotension Measurably Enhance Attention and Memory Functions in Parkinson's Disease
Brief Title: Improved Orthostatic Tolerance = Better Cognitive Function in Parkinson's Disease
Acronym: PaKogOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Andrea Maier, attending physician and investigator, RWTH Aachen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-131
Record Dates: First submitted 2018-12-28; First posted 2019-04-02 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Hypotension, Orthostatic; Parkinson Disease; Autonomic Failure; Cognitive Impairment
MeSH Terms: conditions — Hypotension, Orthostatic; Parkinson Disease; Pure Autonomic Failure; Cognitive Dysfunction | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short_Physiotherapy (Other): one period of physiotherapy (8 weeks)
  Interventions: Other: Physiotherapy
- Long_Physiotherapy (Other): two periods of physiotherapy (à 8 weeks)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Ambulatory leg-muscle oriented physiotherapy (2 x 45 minutes per week for at least 8 weeks) at Aachen University Hospital. Daily protocol of leg muscle training, exercises, sufficient fluid intake of 2liter/day, pressure stockings.

SUMMARY:
Study on orthostatic Hypotension in Parkinson's disease

DETAILED DESCRIPTION:
Orthostatic hypotension (OH) in Parkinson's disease (PD) may not only be related to dizziness or light headedness but to deficits in attention, visual, and verbal memory. Would a successful treatment of OH which includes physiotherapy significantly improve OH and these cognitive deficits? By means of a randomized cross-over trial, we want to measure and compare the effects of OH therapy on orthostatic tolerance, as well as on attention, visuo-spatial working memory, and verbal memory in patients with PD. If confirmed, therapy of orthostatic hypotension would provide a sound and simple approach to improve those cognitive deficits originating from orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's patients
* Diagnostis of OH
* able to perform an ambulatory physiotherapy at Aachen University Hospital.

Exclusion Criteria:

* deep brain stimulation or Pacemaker
* severe psychiatric disease
* severe heart disease
* severe vascular encephalopathy
* dementia
* pregnant or lactating women
* extreme pain or immobility

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure in mmHg | 10months
  Systolic postural blood pressure drop in the interventional Group (Long_Physiotherapy) less than 10mmHg (5-15mmHg) compared to Short_Physiotherapy

SECONDARY OUTCOMES:
Attention in TAP | 10months
  Attention Tasks (TAP) ≥ 20% Change in Long_Physiotherapy
Orthostatic symptoms (Winkler Scale) | 10months
  ≥ 2 points change in Winkler Scale (Sum Score) in Long_Physiotherapy; 10 symptoms must be rated concerning their frequency from 0= never to 4= more than once a day. Sum score from minimum 0 points (no symptoms) to maximum 40 points (all symptoms more than once daily) is interpreted
daytime sleepiness | 10months
  Epworth Sleepiness Scale ≥ 20% Change of Sum Score in Long_Physiotherapy. Sum Score can range from minimum = 0 Points to Maximum = 24points. More points indicate more symptoms. Cut off for daytime sleepiness are10 points

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Maier, Dr. med., Principal Investigator — Universitiy hospital RWTH Aachen, Department of Neurology
Locations (1):
- University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Husch S, Schauermann J, Fimm B, Haubrich C, Reetz K, Schulz JB, Maier A. Effect of strength training on orthostatic hypotension in Parkinson's disease-a pilot study. Clin Auton Res. 2022 Jun;32(3):213-217. doi: 10.1007/s10286-022-00870-5. Epub 2022 Jun 15. No abstract available. PMID 35705801
- See also: Results of the study — https://pubmed.ncbi.nlm.nih.gov/35705801/